CLINICAL TRIAL: NCT01784640
Title: A Phase IB Dose-Escalation Study of Pemetrexed and AUY922 in Previously-Treated Patients With Metastatic Non-Squamous, Non-Small Cell Lung Cancer
Brief Title: Pemetrexed Disodium and Hsp90 Inhibitor AUY922 in Treating Patients With Previously Treated Stage IV Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: Translational Research in Oncology (Other); Novartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12-001489; NCI-2013-00410 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); L-05 (Other: Tanslational Research in Oncology (TRIO))
Record Dates: First submitted 2013-02-05; First posted 2013-02-06 (Estimated); Last update posted 2020-09-03 (Actual); Status verified 2018-04

CONDITIONS: Recurrent Non-small Cell Lung Cancer; Squamous Cell Lung Cancer; Stage IV Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — 5-(2,4-dihydroxy-5-isopropylphenyl)-4-(4-morpholin-4-ylmethylphenyl)isoxazole-3-carboxylic acid ethylamide; Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (Hsp90 inhibitor AUY922, pemetrexed disodium) (Experimental): Patients receive Hsp90 inhibitor AUY922 IV over 60 minutes weekly and pemetrexed disodium IV over 15 minutes every 3 weeks. Courses repeat every 21 days for 6 months in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Hsp90 inhibitor AUY922; Drug: pemetrexed disodium; Other: pharmacological study; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: Hsp90 inhibitor AUY922 — Given IV
  Other Names: AUY922
Drug: pemetrexed disodium — Given IV
  Other Names: ALIMTA; LY231514; MTA
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase I trial studies the side effects and the best dose of Hsp90 inhibitor AUY922 when given together with pemetrexed disodium in treating patients with previously treated stage IV non-small cell lung cancer. Hsp90 inhibitor AUY922 may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as pemetrexed disodium, work in different ways to stop the growth of tumor cell, either by killing the cells or stopping them from dividing. Giving Hsp90 inhibitor AUY922 together with pemetrexed disodium may kill more tumor cells

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Evaluate the safety and tolerability of escalating doses of AUY922 (Hsp90 inhibitor AUY922) when given with pemetrexed (pemetrexed disodium) 500 mg/m^2 in participants with previously-treated stage IV non-squamous, non-small cell lung cancer (NSCLC).

SECONDARY OBJECTIVES:

I. Determine the objective tumor response rate as defined by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria in participants with previously treated non-squamous NSCLC treated with pemetrexed and AUY922.

II. Evaluate the pharmacokinetic profile of pemetrexed and AUY922. III. Evaluate toxicity, including visual toxicity, in participants treated with AUY922 and pemetrexed.

IV. Analyze tumor-tissue biomarkers for potential correlation with response.

OUTLINE: This is a dose-escalation study of Hsp90 inhibitor AUY922.

Patients receive Hsp90 inhibitor AUY922 intravenously (IV) over 60 minutes weekly and pemetrexed disodium IV over 15 minutes every 3 weeks. Courses repeat every 21 days for 6 months in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand the purpose and risks of the study and provide signed and dated informed consent and authorization to use protected health information (PHI) in accordance with national and local subject privacy regulations
* Histologically- or cytologically-confirmed stage IV non-squamous, NSCLC who have progressed after at least one prior line of treatment; in the expansion phase, participants are only eligible if their molecular category has not been fully enrolled (10 participants with epidermal growth factor receptor (EGFR) mutations, 5 participants with anaplastic lymphoma receptor tyrosine kinase (ALK) gene rearrangement, 5 participants with wild type v-Ki-ras2 Kirsten rat sarcoma viral oncogene homolog (KRAS), EGFR and ALK)
* At least one measurable lesion as defined by modified RECIST version 1.1; previously irradiated lesions are not measurable unless the lesion is new or has demonstrated clear progression after radiation
* Last chemotherapy or treatment with another systemic anti-cancer agent must have stopped >= 4 weeks prior to enrollment (or >= 5 half-lives for oral tyrosine-kinase inhibitors or 2 weeks for palliative radiotherapy); participants must have recovered (Common Terminology Criteria for Adverse Events [CTCAE] =< 1 or baseline) from acute toxicities of any previous therapy (with the exception of alopecia)
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2
* Expected survival time of >= 3 months in the opinion of the investigator
* Absolute neutrophil count (ANC) >=1.5 x 10^9/L
* Hemoglobin (Hgb) >= 9 g/dl
* Platelets (plt) >= 100 x 10^9/L
* Potassium within normal limits
* Total calcium (corrected for serum albumin) within normal limits or corrected with supplements
* Magnesium within lower limits or corrected with supplements
* Phosphorus within lower limits or corrected with supplements
* Aspartate aminotransferase (AST)/serum glutamic oxaloacetic transaminase (SGOT) and alanine aminotransferase (ALT)/serum glutamate pyruvate transaminase (SGPT) =< 1.5 x upper limit of normal (ULN)
* AST/SGOT and ALT/SGPT =< 2.5 x upper limit of normal (ULN) if liver metastases are present
* Serum bilirubin =< 1.5 x ULN
* Serum creatinine =< 1.5 x ULN or 24-hour clearance >= 50 ml/min
* Negative serum or urine pregnancy test; the serum pregnancy test must be obtained prior to the first administration of AUY922 (=< 14 days prior to dosing) in all pre-menopausal women and women < 2 years after the onset of menopause
* Ability to provide a formalin-fixed, paraffin-embedded (FFPE) tumor tissue sample containing representative tumor tissue from a previously obtained biopsy/resection that meets specific tissue sample requirements at screening

Exclusion Criteria:

* Unresolved diarrhea >= CTCAE (v4.0) grade 1
* Pregnant or lactating women
* Fertile women of childbearing potential (WCBP) not using (or refusing to use) adequate methods of contraception as agreed on between her and the consenting investigator; male participants not using (or refusing to use) a condom during intercourse
* History of another primary cancer within 3 years prior to enrollment with the exception of curatively treated skin cancer (other than melanoma) or curatively treated cervical carcinoma in-situ
* History of central nervous system (CNS) metastasis; Note: participants without clinical signs and symptoms of CNS involvement are not required to have magnetic resonance imaging (MRI) of the brain; (exception: participants with treated brain metastases who are asymptomatic, not currently on steroid therapy, and clinically stable for >= 2 weeks will be eligible for protocol participation)
* Prior treatment with pemetrexed
* Prior anti-neoplastic treatment with any heat shock protein 90 (HSP90) or histone deacetylase (HDAC) inhibitor compound
* Participants who have undergone any major surgery =< 2 weeks prior to starting study drug or who have not recovered from side effects of such therapy
* Last chemotherapy or treatment with another systemic anti-cancer agent must have stopped >= 4 weeks prior to enrollment (or >= 5 half-lives for oral tyrosine-kinase inhibitors); participants with EGFR mutations and ALK gene rearrangement who have not received a tyrosine kinase inhibitor targeting their molecular abnormality (e.g., erlotinib or crizotinib respectively); participants must have recovered (CTCAE =< 1) from acute toxicities of any previous therapy (with the exception of alopecia)
* Participants who have concurrent or uncontrolled illness that the investigator feels will impede study participation including, but not limited to:

  * Acute or chronic liver disease
  * Acute or chronic renal disease
  * Active or ongoing infection
  * Psychiatric illness/social situations that would limit compliance with study requirements
* Participants with known disorders due to a deficiency in bilirubin glucuronidation (e.g. Gilbert's syndrome)
* Intolerance of Vitamin B12, folic acid or dexamethasone
* Participants with following cardiac criteria:

  * History of long QT syndrome
  * QTcF >= 450 ms during screening electrocardiogram (ECG)
  * History of clinically manifest ischemic heart disease including myocardial infarction, stable or unstable angina pectoris, coronary arteriography or cardiac stress testing/imaging with findings consistent with infarction or clinically significant coronary occlusion ≤ 6 months prior to study start
  * History of heart failure or left ventricular (LV) dysfunction (LV ejection fraction [EF] =< 45%) by multi gated acquisition scan (MUGA) or echocardiogram (ECHO)
  * Clinically significant ECG abnormalities including one or more of the following: left bundle branch block (LBBB), right bundle branch block (RBBB) with left anterior hemiblock (LAHB); ST segment elevations or depressions > 1mm, or 2nd (Mobitz II) or 3rd degree atrioventricular block (AV) block
  * History and presence of atrial fibrillation, atrial flutter or ventricular arrhythmias including ventricular tachycardia or Torsades de pointes
  * Other clinically significant heart disease (e.g. congestive heart failure, uncontrolled hypertension, history of labile hypertension, or history of poor compliance with a hypertensive regimen)
  * Clinically significant resting bradycardia (< 50 beats per minute)
  * Participants who are currently receiving treatment with any medication which has a relative risk or prolonging the QTcF interval or inducing Torsades de pointes (as listed in protocol) and cannot be switched or discontinued to an alternative drug prior to commencing AUY922 dosing
  * Participants who are on a cardiac pacemaker
* Participants unwilling or unable to comply with the protocol
* Participants known to be human immunodeficiency virus (HIV) positive; testing is not required in the absence of clinical signs and symptoms suggesting HIV infection
* Any systemic anti-cancer treatment out of allowed timelines
* Concurrent cytotoxic or immunosuppressive therapy for non-malignant disease (e.g., for rheumatoid arthritis or lupus)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2014-01-31 (Actual); Primary Completion 2018-10-11 (Actual); Study Completion 2018-10-11 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events (AEs) as assessed by National Cancer Institute (NCI) CTCAE version 4.0 | Up to 30 days after completion of study treatment
  Safety will be assessed through tabulation, grading and attribution of serious adverse events (SAEs) and AEs.

SECONDARY OUTCOMES:
Tumor response rate according to RECIST version 1.1 | Up to 30 days after completion of study treatment
  The proportion of ever achieving a clinical response will be estimated and constructed with an exact one-sided 90% confidence interval to identify the likely range for the underlying tumor response rate. Clinical response will be correlated with biomarkers using a variety of analytic techniques.

CONTACTS AND LOCATIONS:
Overall Officials: Edward Garon, Principal Investigator — Jonsson Comprehensive Cancer Center
Locations (1):
- Jonsson Comprehensive Cancer Center, Los Angeles, California, United States